CLINICAL TRIAL: NCT04870671
Title: Project ADHERE: Clinical Proof-of-Concept of a Tenofovir (TFV) Aptamer-Based Biosensor for Determining Adherence Using Different Dosing Regimens of Disoproxil Fumarate/Emtricitabine (TDF/FTC)
Brief Title: Project ADHERE: Clinical Proof-of-Concept of a Tenofovir (TFV) Aptamer-Based Biosensor
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Eastern Virginia Medical School (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Terry Jacot, Research Assistant Professor, Eastern Virginia Medical School
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 19-08-FB-0195; 5R21AI145809-02 (NIH)
Record Dates: First submitted 2021-04-23; First posted 2021-05-03 (Actual); Results first posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: HIV/AIDS; Adherence, Medication; Drug Use
Keywords: HIV PrEP; biosensor; tenofovir
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Medication Adherence | interventions — Tenofovir; Emtricitabine; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Intervention Model Description: Women will be randomized into one of two groups: high adherence (7 pills/week) and how adherence (3 pills/week)
Who Masked: Outcomes Assessor
Masking Description: When measuring TFV levels in the biological fluids, the outcomes assessor in the laboratory will not know whether the samples are from the high or low adherence group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- High Adherence (Experimental): TDF/FTC (300/200 mg), 7 pills/week. Total of 14 pills
  Interventions: Drug: Tenofovir Disoproxil Fumarate/Emtricitabine (TDF/FTC)
- Low Adherence (Experimental): TDF/FTC (300/2200 mg), 3 pills/week. Total of 6 pills
  Interventions: Drug: Tenofovir Disoproxil Fumarate/Emtricitabine (TDF/FTC)

INTERVENTIONS:
Drug: Tenofovir Disoproxil Fumarate/Emtricitabine (TDF/FTC) — Women will take 1 pill orally according the dosing regimen of the arm to which they are assigned
  Other Names: Truvada

SUMMARY:
Truvada®, an oral pill comprised of two anti-retroviral compounds, emtricitabine (FTC) and tenofovir disoproxil fumarate (TDF), is currently the only drug combination approved for pre-exposure prophylaxis (PrEP) in women exposed to high HIV risk through vaginal acquisition. Adherence to the one pill per day regimen is crucial for its effectiveness in reducing the risk of acquiring HIV. Currently, there is no available point of care diagnostic test to quickly measure blood levels of tenofovir in the clinic. This study will determine whether a tenofovir (TFV) aptamer-based biosensor (aptasensor) can detect TFV in biological fluids from women randomized to different dosing regimens representing high and low adherence.

DETAILED DESCRIPTION:
Project ADHERE is a pilot, prospective, randomized study which will screen approximately 20 healthy, non-pregnant, HIV negative, premenopausal women (aged 18-50) at Eastern Virginia Medical School (EVMS) who are not at risk of pregnancy and are at low risk for sexually transmitted infections (STIs) in order to have approximately 14 women complete all study visits. The women will be randomized to one of two different dosing regimens of Truvada for up to 14 days. The low adherence cohort will take a total of 3 Truvada pills per week while the high adherence cohort will be assigned to take daily dosing, 7 pills per week. At screening (visit 1), we will screen women for HIV-1 and perform STI tests and serum screening for Hepatitis B and creatinine clearance prior to commencing oral PrEP, consistent with oral PrEP initiation guidelines. After screening labs return, they will come to the clinic for visit 2 when baseline blood, urine, and vaginal fluid will be collected, randomize participants to the dosing regimen, watch the participants ingest the first dose, and then direct to them to take subsequent doses in their homes. Reminder text messages will be sent to the participants to facilitate doses being taken at the same time of day upon which they will text message the coordinator after ingesting the pill. Participants will return 24 hours, 7 days, and 14 days after visit 2 for pre-dose collection of blood, urine, and vaginal fluid samples (visits 3, 4, and 5, respectively). For all visits, participants will not to take the next prescribed dose before coming to the clinic. Once samples are collected, participants will ingest the next scheduled pill. However, for the high adherence regimen, the women will take their last dose on day 14 and then come to the clinic 24 hours later on day 15 for collection of samples. Regardless of regimen, sample collection will take place no earlier than 24 hours after last dosing to prevent white coat effects. Samples will be brought to the laboratory for processing and eventual measurement of TFV levels by the TFV aptasensor. Aliquots of plasma and urine will also be analyzed by Liquid Chromatography-Tandem Mass Spectrometry (LC-MS/MS) so sensitivity and specificity of the aptasensor can be determined. The ability of the TFV aptasensor to distinguish levels associated with high and low adherence will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 50 years, inclusive
* General good health (by volunteer history and per investigator judgment) without any clinically significant systemic disease (including, but not limited to significant liver disease/hepatitis, gastrointestinal disease, kidney disease, thyroid disease, osteoporosis or bone disease, and diabetes) and with an intact gastrointestinal tract, uterus and cervix.
* Estimated calculated creatinine clearance (eCcr) of at least 80 mL/min
* Body Mass Index (BMI) of ≥18 and <35kg/m2; and a total body weight >45 kg (99.2 lbs)
* Willing to give voluntary consent and sign an informed consent form
* Willing and able to comply with protocol requirements, including swallowing tablets
* Must be protected from pregnancy by:

  1. Condoms
  2. Hormonal contraceptives
  3. Copper or Levonorgestrel intrauterine device (IUD)
  4. Sterilization of either partner
  5. Heterosexual abstinence
  6. Same sex relationship
* If in a relationship, must be in a mutually monogamous relationship with a partner who is not known to be HIV positive and has no known risk of STIs

Exclusion Criteria:

* Currently pregnant
* Currently breastfeeding or planning to breastfeed during the course of the study
* In the last three months, diagnosed with or treated for any STI
* Positive test for HIV, or Hepatitis B surface antigen (HBsAg)
* Systemic use in the last two weeks or anticipated use during the study of any of the following: antiretrovirals (e.g. Viread®, Atripla®, Emtriva®, or Complera®), or drugs that may interact with TFV (e.g., protease inhibitors, anticonvulsants, antimycobacterials, St. John's Wort).
* Participation in any other investigational trial with use of a drug/device within the last 30 days or planned participation in any other investigational trial with use of a drug/device during the study
* Grade 2 or higher laboratory abnormality, per the 2014 update of the Division of AIDS, National Institute of Allergy and Infectious Disease (DAIDS) Table for Grading the Severity of Adverse Events, or clinically significant laboratory abnormality as determined by the clinician
* Abnormal finding on laboratory or physical examination or a social or medical condition in the volunteer which, in the opinion of the investigator, would make participation in the study unsafe or would complicate interpretation of data

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 14 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terry A Jacot, PhD, Principal Investigator — Eastern Virginia Medical School; Andrea R Thurman, MD, Principal Investigator — Eastern Virginia Medical School
Locations (1):
- Clinical Research Center, Eastern Virginia Medical School, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ruscito A, DeRosa MC. Small-Molecule Binding Aptamers: Selection Strategies, Characterization, and Applications. Front Chem. 2016 May 10;4:14. doi: 10.3389/fchem.2016.00014. eCollection 2016. PMID 27242994
- [Background] Hendrix CW, Andrade A, Bumpus NN, Kashuba AD, Marzinke MA, Moore A, Anderson PL, Bushman LR, Fuchs EJ, Wiggins I, Radebaugh C, Prince HA, Bakshi RP, Wang R, Richardson P, Shieh E, McKinstry L, Li X, Donnell D, Elharrar V, Mayer KH, Patterson KB. Dose Frequency Ranging Pharmacokinetic Study of Tenofovir-Emtricitabine After Directly Observed Dosing in Healthy Volunteers to Establish Adherence Benchmarks (HPTN 066). AIDS Res Hum Retroviruses. 2016 Jan;32(1):32-43. doi: 10.1089/AID.2015.0182. Epub 2015 Oct 15. PMID 26414912
- [Background] Donnell D, Baeten JM, Bumpus NN, Brantley J, Bangsberg DR, Haberer JE, Mujugira A, Mugo N, Ndase P, Hendrix C, Celum C. HIV protective efficacy and correlates of tenofovir blood concentrations in a clinical trial of PrEP for HIV prevention. J Acquir Immune Defic Syndr. 2014 Jul 1;66(3):340-8. doi: 10.1097/QAI.0000000000000172. PMID 24784763

RESULTS

PARTICIPANT FLOW:
Groups:
- High Adherence: Tenofovir Disoproxil Fumarate/Emtricitabine (TDF/FTC) (300/200 mg), 7 pills/week. Total of 14 pills
  TDF/FTC: Women will take 1 pill orally according the dosing regimen of the arm to which they are assigned
- Low Adherence: Tenofovir Disoproxil Fumarate/Emtricitabine (TDF/FTC) (300/2200 mg), 3 pills/week. Total of 6 pills
  TDF/FTC: Women will take 1 pill orally according the dosing regimen of the arm to which they are assigned
Period: Overall Study
Arm/Group | High Adherence | Low Adherence
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The participants served as their own baseline controls.
Groups:
- Total: Total of all reporting groups
Arm/Group | High Adherence | Low Adherence | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 14
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.1 (10.6) | 37.7 (7.8) | 38.9 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 6 | 7 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 14
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 31.3 (7) | 32.4 (11.8) | 31.8 (9.3)
Creatinine Clearance [Mean (Standard Deviation); unit: mL/min] | 157.2 (48.3) | 169 (77.9) | 163.1 (62.6)

OUTCOME MEASURES:

1. Primary Outcome: Baseline TFV (Tenofovir) Levels in Plasma
Description: TFV levels will be measured by the TFV aptasensor and compared to Liquid Chromatography with Tandem Mass Spectrometry (LC-MS/MS) values
Time Frame: Baseline (pre-dose)
Population: The development of the aptasensor did not reach the target endpoint of detecting TFV in human plasma samples
Groups:
- High Adherence: TDF/FTC (300/200 mg), 7 pills/week. Total of 14 pills
  Tenofovir Disoproxil Fumarate: Women will take 1 pill orally according the dosing regimen of the arm to which they are assigned
- Low Adherence: TDF/FTC (300/2200 mg), 3 pills/week. Total of 6 pills
  Tenofovir Disoproxil Fumarate: Women will take 1 pill orally according the dosing regimen of the arm to which they are assigned
Arm/Group | High Adherence | Low Adherence
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Levels of TFV in Plasma After Different Lengths of Time Post-first Dose
Description: TFV levels will be measured by the TFV aptasensor and compared to LC-MS/MS values
Time Frame: 1 day
Population: The development of the aptasensor did not reach the target of detecting TFV in human plasma samples
Arm/Group | High Adherence | Low Adherence
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Levels of TFV in Plasma After Different Lengths of Time Post-first Dose
Description: TFV levels will be measured by the TFV aptasensor and compared to LC-MS/MS values
Time Frame: 7 days
Population: The development of the aptasensor did not reach the target of detecting TFV in human plasma samples
Arm/Group | High Adherence | Low Adherence
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Levels of TFV in Plasma After Different Lengths of Time Post-first Dose
Description: TFV levels will be measured by the TFV aptasensor and compared to LC-MS/MS values
Time Frame: 14 days
Population: The development of the aptasensor did not reach the target of detecting TFV in human plasma samples.
Arm/Group | High Adherence | Low Adherence
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | High Adherence | Low Adherence
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 2/7 | 2/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Adherence (N=7) | Low Adherence (N=7)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (General disorders) | 1 (1) | 1 (1)
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
increased appetite (General disorders) | 1 (1) | 0 (0)
headache (General disorders) | 1 (1) | 0 (0)
Allergies (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The project was successful in developing an aptasensor that could detect 1-30 nanomolar (nM) TFV in saline. However, the electrode configuration could not detect TFV in plasma due to interfering signals generated by the proteins present in the sample. Therefore, the aptasensor needs optimization before it can successfully be tested against the clinical samples of this clinical trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-29): https://cdn.clinicaltrials.gov/large-docs/71/NCT04870671/Prot_SAP_000.pdf